CLINICAL TRIAL: NCT06205927
Title: Randomized Study of Carbon Ion Boost in Hypoxic Lesions Identified by 18F-Misonidazole PET/CT in Patients With Non-Small Cell Lung Cancer
Brief Title: Randomized Study of Carbon Ion Boost in Hypoxic Lesions for Locally Advanced Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jian Chen (Other)
Responsible Party: Sponsor-Investigator, Jian Chen, Clinical Professor, Shanghai Proton and Heavy Ion Center
Organization: Shanghai Proton and Heavy Ion Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPHIC-TR-THLC2023-02
Record Dates: First submitted 2023-12-17; First posted 2024-01-16 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Non-small Cell Lung Cancer
Keywords: 18Fluoro-misonidazole, hypoxia, particle therapy, carbon-ion radiotherapy, non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard treatment arm (Active Comparator): The standard treatment arm will receive carbon ion beam radiotherapy of 77Gy (RBE equivalent) per 22 fractions for gross tumor volume.
  Interventions: Radiation: Standard carbon ion beam radiotherapy
- Boost arm (Experimental): Boost arm will receive 77Gy (RBE equivalent) per 22 fractions for gross tumor volume and a simultaneously dose boost of 83.6Gy (RBE equivalent) per 22 fractions for hypoxic lesions detected by 18F-Misonidazole PET/CT
  Interventions: Radiation: Carbon ion beam radiotherapy simultaneously dose boost

INTERVENTIONS:
Radiation: Standard carbon ion beam radiotherapy — The standard treatment arm will receive carbon ion beam radiotherapy of 77Gy (RBE equivalent) per 22 fractions for gross tumor volume.
  Arms: Standard treatment arm
Radiation: Carbon ion beam radiotherapy simultaneously dose boost — The hypoxic lesions dose boost arm will receive 77Gy (RBE equivalent) per 22 fractions for gross tumor volume and a simultaneously dose boost of 83.6Gy (RBE equivalent) per 22 fractions for hypoxic lesions detected by 18F-Misonidazole PET/CT.
  Arms: Boost arm

SUMMARY:
The goal of this randomized clinical trial is to learn about if carbon ion radiotherapy dose boost in hypoxia lesions detected by 18F-Misonidazole PET/CT could improve clinical outcomes in locally advanced non-small cell lung cancer patients compared with standard treatment protocol in our center. The patients will be randomly divided into two arms: standard treatment arm and hypoxic lesions dose boost arm. The standard treatment arm will receive carbon ion beam radiotherapy of 77Gy (RBE equivalent) per 22 fractions for gross tumor volume. The hypoxic lesions dose boost arm will receive 77Gy (RBE equivalent) per 22 fractions for gross tumor volume and a simultaneously dose boost of 83.6Gy (RBE equivalent) per 22 fractions for hypoxic lesions detected by 18F-Misonidazole PET/CT.

Researchers will compare the local progression-free survival of two groups (primary endpoint), progression-free survival (secondary endpoint), overall survival (secondary endpoint), response rate (secondary endpoint), factional hypoxia volume (FHV) reduction rate (secondary endpoint) and toxicities (secondary endpoint).

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 80.
* ECOG general status score of 0-2 .
* Primary non-small cell lung cancer (NSCLC) confirmed by histology or cytological pathology, stage IIIa-IIIc (AJCC/UICC 8th edition). Largest diameter of primary tumor ≥ 4cm before carbon ion radiotherapy.
* Medically inoperable, or patient refuses surgery.
* Adequate organ function: 1). Blood function: absolute neutrophil count (ANC) ≥1.5 x 109/L, platelet count ≥80 x 109/L, hemoglobin ≥9 g/dL 2). Lung function: FEV1>25%, DLCO>25% 3). Cardiac function: no serious pulmonary hypertension, cardiovascular and cerebrovascular diseases, peripheral vascular diseases, serious chronic heart disease and other complications that may affect radiotherapy.4). Adequate liver function: total bilirubin <1.5 times the upper limit of normal value, and AST, ALT<2 times the upper limit of normal value. 5). Adequate renal function: serum creatinine ≤1.5 times the upper limit of normal or calculated creatinine clearance ≥50 ml /min, and urinary protein <2+. Patients with a baseline urinary protein level of 2+ or more should have a 24-hour urine collection and evidence of a 24-hour urinary protein level of 1g or less.
* Sign the informed consent.

Exclusion Criteria:

* Patients with squamous cell carcinoma treated with bevacizumab before radiotherapy.
* Patient fails to comply with the treatment protocol.
* Complicated with other malignant tumors that have not been controlled.
* Patient whose particle radiotherapy plan cannot meet the minimum target dose coverage and dose volume limitation requirements, or cannot meet the dose constrains of normal tissue or organs.
* Chest radiation therapy or radioactive particle implantation history.
* Cardiac pacemakers or other internal metal prosthesis implants that may be affected by high-energy radiation or may affect the dose distribution to the radiation target area.
* Pregnancy (confirmed by serum or urine β-HCG test) or lactation period.
* HIV positive. Hepatitis virus replication phase, need to receive antiviral therapy, but because of concomitant disease cannot receive antiviral therapy. Active stage of syphilis.
* A history of mental illness may hinder the completion of treatment.
* With serious comorbidity that may interfere with radiotherapy, including: (a) Acute infectious diseases or acute active phase of chronic infection. b) Unstable angina pectoris, congestive heart failure, myocardial infarction that has been hospitalized in the past 6 months. c) Exacerbations of chronic obstructive pulmonary disease or other respiratory conditions requiring hospitalization. d) Severely impaired immune function. e) Diseases with excessive sensitivity to radiation such as ataxia telangiectasia. f) Other diseases that may affect particle radiotherapy.
* Other circumstances that the physician considers inappropriate to participate in clinical study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2023-12-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Local progression-free survival | From date of radiotherapy started until the date of first documented local disease progression, assessed up to 100 months
  Local progression-free survival was defined from the start of carbon ion radiotherapy till the date of local progression or the last follow-up

SECONDARY OUTCOMES:
Disease progression-free survival rate | From date of radiotherapy started until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Disease progression-free survival rate was defined from the start of carbon ion radiotherapy till the date of disease progression at any site or death, or the last follow up
Overall survival rate | From date of radiotherapy started until the date of death from any cause, assessed up to 100 months
  Overall survival rate was defined from the start of carbon ion radiotherapy till the date of death or the last follow-up
Overall response rate | From date of radiotherapy started until 6 months after first radiotherapy
  Proportion of complete response and partial response in all patients
Change of fractional hypoxia volume | From date of radiotherapy started until 1 month after first radiotherapy
  The hypoxia volume of the hypoxia-positive region of interested was defined as the sum of pixels with a tumor muscle rate ≥1.4. The FHV, defined as the HV-to-gross tumour volume ratio. The FHV before and after carbon ion radiotherapy within 1 month will be recorded.
Incidence of Treatment-induced Adverse Events | From date of radiotherapy started, every 3-4 months within the first 2 years, every 6 months between years 3 and 5, and annually thereafter, assessed up to 100 months
  Treatment-induced toxicities were scored using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 and EORTC/RTOG criteria, for events observed after the first dose of irradiation. Toxicities occurred 90 or more days after the completion of CIRT were defined as late toxicities.

CONTACTS AND LOCATIONS:
Overall Officials: Jingfang Mao, PHD, Study Chair — Shanghai Proton and Heavy Ion Center
Locations (1):
- Shanghai Proton and Heavy Ion Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided